CLINICAL TRIAL: NCT00456976
Title: Efficacy of Selegiline Augmentation of Antipsychotic Medication to Treat Negative Symptoms in Inpatients With Chronic Schizophrenia
Brief Title: Efficacy of Selegiline in Negative Symptoms of Schizophrenia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tabriz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8514; tums
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2008-07-23 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
Keywords: Seligiline; Negative symptoms; Schizopherenia
MeSH Terms: conditions — Schizophrenia | interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Selegiline

SUMMARY:
Antipsychotic drugs are effective in treating the positive symptoms of schizophrenia; however their efficacy in treating negative symptoms is limited. This study wants to evaluate efficacy of selegiline augmentation of antipsychotic medication to treat negative symptoms in inpatients with chronic schizophrenia. With randomized clinical trial two groups of patients will select to receive selegiline or placebo.

Primary end point is decreasing in negative symptoms in case group. Inclusion criteria : 1- Patients with moderate to severe negative symptoms 2- Patients with at least one year antipsychotic drug therapy, at the current dose >= 1 month. 3- No other psychotropic drugs during past month. Exclusion criteria: 1- Severe major depressive disorder, substance abuse, severe positive symptoms of schizophrenia, Treatment of MDD with antidepressant drugs during past month.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe negative symptoms
* Patients with at least one year antipsychotic drug therapy, at the current dose >= 1 month.
* No other psychotropic drugs during past month

Exclusion Criteria:

* Severe major depressive disorder
* Substance abuse
* Severe positive symptoms of schizophrenia
* Treatment of MDD with antidepressant drugs during past month.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2007-04; Study Completion 2007-09

PRIMARY OUTCOMES:
decreasing in negative symptoms in case group

CONTACTS AND LOCATIONS:
Overall Officials: Fatemeh Ranjbar Kouchaksaraei, Assistant Professor, Study Chair — Tabriz University of Medical Sciences
Locations (1):
- Razi university hospital, Tabriz, East Azerbaijan Province, Iran